CLINICAL TRIAL: NCT01708681
Title: Ability of a Lean Seafood Diet to Modulate Postprandial Metabolism in Human-beings - a Controlled Intervention Study With Cross-over Design
Brief Title: Lean Seafood Intake and Postprandial Metabolism
Acronym: LeSIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Nutrition and Seafood Research, Norway (Other Government)
Collaborators: The Research Council of Norway (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: NIFES-001; 2012/1084/REK vest (Other Grant/Funding Number: NRC-200515/I30)
Record Dates: First submitted 2012-10-11; First posted 2012-10-17 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Hyperlipidemias; Nutritional and Metabolic Diseases; Nutrition Disorders; Metabolic Diseases; Glucose Metabolism Disorders
Keywords: Seafood; Meat; Egg; Milk; Postprandial lipid metabolism; Postprandial glucose metabolism; Triglycerides; Cholesterol; Postprandial incretins; Postprandial hormones
MeSH Terms: conditions — Hyperlipidemias; Nutritional and Metabolic Diseases; Nutrition Disorders; Metabolic Diseases; Glucose Metabolism Disorders | interventions — Meat; Eggs; Milk

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Lean seafood (Experimental): Cross-over design, half of the subject will receive lean seafood in study period I and the other half in study period II
  Interventions: Dietary Supplement: Lean seafood; Dietary Supplement: Meat, egg, milk
- Meat, egg, milk (Active Comparator): Cross-over design, half of the subject will receive meat, egg, milk in study period I and the other half in study period II
  Interventions: Dietary Supplement: Lean seafood; Dietary Supplement: Meat, egg, milk

INTERVENTIONS:
Dietary Supplement: Lean seafood
Dietary Supplement: Meat, egg, milk

SUMMARY:
Despite numerous studies of meal components in humans, little is still known about how different meals influence on metabolism. The purpose of this study is to a gain knowledge of how a balanced test meal with either lean seafood (example:cod) or meat as the main protein source will:

1. affect the postprandial metabolism acutely (test-meal at beginning of the study)
2. affect the postprandial metabolism after 4 weeks controlled intervention (test meal at end of intervention period)
3. affect gut microbiota composition

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Caucasian

Exclusion Criteria:

* Smoking
* Diabetes
* Hysterectomy
* Abnormal bleeding last 6 months
* Use of medication that affects lipid and glucose metabolism
* Large (>10%) alteration in body-weight the last 6 months
* Chronic, metabolic or acute disease or major surgery within last 3 months
* Dietary incompatibility with calcium supplementation and/ or seafood consumption (allergy, intolerance, dislike)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2012-10; Primary Completion 2013-05 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Postprandial lipid measurement | Change from baseline at 4 weeks

SECONDARY OUTCOMES:
Postprandial glucose measurement | Change from baseline at 4 weeks

OTHER OUTCOMES:
Postprandial metabolomic measurement | Change from baseline at 4 weeks
Gut microbiota composition | Change from baseline at 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bjørn Liaset, Dr, Principal Investigator — NIFES
Locations (1):
- National Institute of Nutrition and Seafood Research, Bergen, Norway

REFERENCES:
- [Derived] Aadland EK, Graff IE, Lavigne C, Eng O, Paquette M, Holthe A, Mellgren G, Madsen L, Jacques H, Liaset B. Lean Seafood Intake Reduces Postprandial C-peptide and Lactate Concentrations in Healthy Adults in a Randomized Controlled Trial with a Crossover Design. J Nutr. 2016 May;146(5):1027-34. doi: 10.3945/jn.115.229278. Epub 2016 Apr 20. PMID 27099232
- [Derived] Aadland EK, Lavigne C, Graff IE, Eng O, Paquette M, Holthe A, Mellgren G, Jacques H, Liaset B. Lean-seafood intake reduces cardiovascular lipid risk factors in healthy subjects: results from a randomized controlled trial with a crossover design. Am J Clin Nutr. 2015 Sep;102(3):582-92. doi: 10.3945/ajcn.115.112086. Epub 2015 Jul 29. PMID 26224298
- See also: Related Info — http://www.nifes.no